CLINICAL TRIAL: NCT06655662
Title: An Open, Multi-center, Phase I Clinical Study on the Safety and Efficacy of HGI-001 Injection in Patients with Transfusion-Dependent Β-Thalassemia.
Brief Title: Evaluating Safety and Efficacy of Lentiviral-transduced CD34+ HSCs in Β-thalassaemia Patients.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Shenzhen Hemogen (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HGI-001C04
Record Dates: First submitted 2024-10-18; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Β-thalassemia
Keywords: β-thalassemia; Thalassemia; Genetic Diseases, Inborn; Hemoglobinopathies; Hematologic Diseases; Anemia; Anemia, Hemolytic; Anemia, Hemolytic, Congenital
MeSH Terms: conditions — Thalassemia; Genetic Diseases, Inborn; Hemoglobinopathies; Hematologic Diseases; Anemia; Anemia, Hemolytic; Anemia, Hemolytic, Congenital

STUDY DESIGN:
Intervention Model Description: This phase 1 study employs a single-group, open-label design to evaluate the safety and preliminary efficacy of a gene therapy product. It is anticipated that 8 participants will be enrolled to receive a single administration of the investigational gene therapy. The primary focus will be on monitoring participants for adverse events and assessing the product's safety profile and potential therapeutic benefits.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- β-globin-restored autologous hematopoietic stem cells modified with LentiHBBT87Q (Experimental): This arm involves the transduction of autologous hematopoietic stem cells with a lentiviral vector carrying the β-globin gene modified with LentiHBBT87Q. Subjects aged 6-35 years with transfusion-dependent β-thalassaemia will receive a infusion of these modified stem cells.
  Interventions: Other: β-globin restored autologous hematopoietic stem cells

INTERVENTIONS:
Other: β-globin restored autologous hematopoietic stem cells — Eight transfusion-dependent β-thalassaemia subjects aged 6-35 years will be reinfused with β-globin restored autologous hematopoietic stem cells modified with LentiHBBT87Q

SUMMARY:
This is a single-arm, open label, multi-center, single-dose Phase 1 clinical trial in subjects with transfusion dependent β-thalassaemia. The study aims to evaluate the safety and efficacy of autologous lentiviral-transduced CD34+ human hematopoietic stem cells (hHSCs) using the gene therapy product HGI-001.

DETAILED DESCRIPTION:
The investigators will recruit transfusion-dependent β-thalassaemia patients and collect their autologous hematopoietic stem cells, which will be modified with the LentiHBBT87Q system to restore β-globin expression. After conditioning, the autologous hematopoietic stem cells with restored β-globin will be reinfused to the patients and followed up for two years to collect data.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 6-35 years (inclusive), ICF can be provided by the patient and/or legal guardian;
2. Definitively diagnosed with severe TDT without genotype restriction (excluding patients with coexisting α-thalassemia), and a valid test report can be provided;
3. Average transfusion volume > 100 mL/kg/year or transfusion frequency > 8 times/year within 2 years prior to enrollment；
4. At least 3 months of full volume transfusion (verification of blood transfusion records can be provided) prior to screening, and Hb is maintained at ≥ 9.0 g/dL;
5. Serum ferritin level less than 5000μg/L, with moderate or lower iron overload in the heart and liver as indicated by magnetic resonance imaging (MRI T2*), specifically liver MRI T2* greater than 1.4ms and cardiac MRI T2* greater than 10ms;
6. Acceptable organ functions (including heart, liver, kidney, lung and coagulation functions), stable disease condition, and suitable for busulfan pre-treatment and hematopoietic stem cell (HSC) transplantation as judged by the investigator;
7. Meets follow-up requirements, adheres to treatment arrangements, and is able to return to the hospital regularly to undergo various examinations within 2 years after reinfusion of HGI-001 injection.

Exclusion Criteria:

1. Patients with fully HLA-matched donors;
2. Having previously received gene therapy, gene editing therapy, or allogeneic hematopoietic stem cell transplantation;
3. Uncorrected bleeding disorder;
4. Uncontrolled epilepsy and mental illness;
5. Within the past 3 months prior to enrollment, the use of Luspatercept, Hydroxyurea, Ruxolitinib, Thalidomide, Decitabine, or Ara-c has been administered；
6. Psychoactive substance abuse, drug or alcohol abuse within 6 months prior to enrollment;
7. Patients with pulmonary hypertension who have not been given effective intervention;
8. Positive for anti-RBC antibodies in antibody screening;
9. Hepatitis B surface antigen (HBsAg) is positive and the HBV DNA copy number is greater than the upper limit of the normal value of the detection unit (those who are negative do not need to test for HBV DNA copy number), antibodies to Hepatitis C virus (HCV) are positive, antibodies to Human Immunodeficiency Virus (HIV) are positive, or antibodies to Treponema pallidum (TP-Ab) are positive (subjects who are positive due to vaccination are eligible for enrollment). Additionally, the results of Hepatitis B Virus (HBV) DNA testing, Hepatitis C Virus (HCV) RNA testing, Cytomegalovirus DNA testing, and Epstein-Barr Virus (EBV) DNA testing are abnormal；
10. Have or have had malignant tumors or myeloproliferative diseases or immunodeficiency disorders or autoimmune diseases;
11. Have a first-degree relative with a history of or suspected hereditary cancer (including but not limited to hereditary breast and ovarian cancer, nonpolyposis colorectal cancer, and adenomatous polyposis);
12. Severe bacterial, viral, fungal or parasitic infection;
13. Other illnesses which render the subject unsuitable for participation (e.g., severe liver, kidney or heart disease); Definition of severe liver and kidney disease: a. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), or total bilirubin > 3 × ULN; b. Liver magnetic resonance imaging (MRI) indicates significant cirrhosis; c. Liver biopsy indicates cirrhosis, severe fibrosis or active hepatitis (liver biopsy is only performed when liver MRI indicates active hepatitis and significant fibrosis without evidence for cirrhosis); d. Creatinine clearance <60 mL/(min·1.73m^2);
14. WBC < 3 × 10^9/L and/or PLT < 100 × 10^9/L;
15. Has diabetes, abnormal thyroid functions or other endocrine disorder;
16. Participated in other interventional clinical studies within 4 weeks before the trial;
17. Poor adherence or other conditions that renders the subject unsuitable for participation as judged by the investigator.

Ages: 6 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2024-06-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Transfusion Independence (TI) Rate | 0-24 Months
  Percent of subjects who achieve transfusion independence, defined as not requiring transfusion for at least 12 consecutive months post-HGI-001 injection, with a weighted average Hb of ≥ 9.0 g/dL. Calculated from the point hemoglobin reaches ≥9 g/dL and no transfusions have occurred in the last 60 days.
Incidence and Severity of Adverse Events (AEs) Related to Transplantation | 0-24 Months
  Number and percentage of adverse events related to transplantation, summarized according to NCI CTCAE 5.0.
Incidence of Serious Adverse Events (SAEs) Related to Transplantation | 0-24 Months
  Number of serious adverse events related to transplantation, summarized according to NCI CTCAE 5.0.
Overall Survival Rate During the Clinical Trial | 0-24 Months
  Number of patients alive throughout the entire trial period.
Percentage of Negative Replicating Lentivirus Test Post-HGI-001 Injection | 0-24 Months
  The percentage of participants with negative results for replicating lentivirus in the 24 months following HGI-001 injection.
Number of Participants with Normal Clonal Variations Post-Transplant | 0-24 Months
  Evaluation of the percentage of participants who do not exhibit abnormal clonal proliferation and maintain polyclonal engraftment following transplantation.
Number of Participants Experiencing Transplantation-related Fatal and Disabling Events Within 100 Days Post-transplantation | 0-100Days
  The number of participants who experience transplantation-related fatal and disabling events within 100 days after transplantation will be recorded and summarized.
Number of Patients with Abnormal Hematology and Bone Marrow Cytology Post-Reinfusion | 0-24 Months
  Number of patients exhibiting abnormal hematology and bone marrow cytology findings within 24 months after reinfusion, and the percentage of patients with abnormal RBC proliferation.

SECONDARY OUTCOMES:
Percentage of Subjects Achieving Transfusion Cessation for Over 6 Months Post-HGI-001 Injection | 0-24 Months
  Percent of subjects who do not require transfusion for at least 6 consecutive months after reinfusion of HGI-001 injection
Percentage of Subjects with Successful HSC Engraftment | 1 month
  Percentage of subjects meeting criteria for successful engraftment, defined as an absolute neutrophil count > 0.5 × 10^9/L for 3 consecutive days and a platelet count maintained at > 20 × 10^9/L for 7 consecutive days without platelet transfusion.
Percentage Change in Annual Transfusion Volume or Frequency | 0-24 Months
  Percentage change in average annual transfusion volume or frequency from baseline.
Transfusion Improvement Rate | 0-24 Months
  Percentage of subjects with a decrease of 30% or more in the average annual transfusion volume or frequency (0-12 months, 12-24 months) from baseline after reinfusion of HGI-001 injection.
Change in Vector Copy Number (VCN) Post-Transplantation | 0-24 Months
  The change in vector copy number (VCN) from the baseline measurement at the time of transplantation to 24 months post-transplantation, as assessed by quantitative PCR.
Change in Exogenous Adult Hemoglobin HbAT87Q Expression Levels Post-Transplantation | 0-24 Months
  The change in expression levels of exogenous adult hemoglobin HbAT87Q from baseline to 24 months post-transplantation, calculated using high-performance liquid chromatography (HPLC) in conjunction with the ratio of HbA to total hemoglobin.
Changes in Cardiac and Liver Iron Load Post-HGI-001 Infusion | 0-24 Months
  Assessment of the changes in cardiac and liver iron load as measured by MRI T2* imaging following the reinfusion of HGI-001 injection.
Time to and Duration of Transfusion Independence in Subjects Post-HGI-001 Infusion | 0-24 Months
  Time from Day 0 to achievement of transfusion independence (TI) and the duration of maintaining TI; average total hemoglobin (Hb) and HbAT87Q levels during the TI period.
Change in Serum Ferritin Levels Post-HGI-001 Infusion | 0-24 Months
  The change in serum ferritin levels following the reinfusion of HGI-001 injection.

CONTACTS AND LOCATIONS:
Overall Officials: Chao Liu, PHD, Principal Investigator — Shenzhen Hemogen; Sixi Liu, Professor, Principal Investigator — Shenzhen Children's Hospital; Yongrong Lai, Professor, Principal Investigator — First Affiliated Hospital of Guangxi Medical University
Locations (3):
- China (3):
  - Guangxi Medical University First Affiliated Hospital, Guangxi
  - Shenzhen Children's Hospital, Shenzhen
  - Shenzhen University General Hospital, Shenzhen

IPD SHARING:
Plan to Share IPD: No